CLINICAL TRIAL: NCT04480112
Title: Impact of Frequent Social Interaction Through Communication Technologies in the Cognitive Status of Socially-isolated Older Adults With and Without Cognitive Impairment
Brief Title: Impact of Covid-19 on Frequent Social Interaction Through Communication Technologies in the Cognitive Status of Socially-isolated Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H-26786
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Memory Disorders; Alzheimer Disease; Mild Cognitive Impairment
Keywords: Social Isolation; Cognition; Misinformation
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease; Cognitive Dysfunction; Social Isolation; Communication

STUDY DESIGN:
Intervention Model Description: The investigators will employ an AB/BA crossover design (2-sequence, 2-period, 2-treatment design) where A will be the intervention phase and B will be the passive control phase. Each period will have a duration of 1 month. Assessment of the primary outcome will be done at the end of each period. Since this is a study of a behavioral intervention, 4-week washout period will suffice to observe an acute change in cognitive performance without significant carryover effects.
  To avoid imbalance among groups, randomization will be stratified by cognitive syndrome diagnosis (healthy older adult, mild cognitive impairment and mild dementia). Participants will be randomized to the treatment sequences using a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: Trial investigators and outcome assessors will be blind to the treatment randomization and allocation..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Intervention (Experimental): Participants in Group A will receive an intervention designed to provide participants with more social interaction during a time of social distancing and highly limited in-person social interactions
  Interventions: Behavioral: Technology based social interactions
- Group B Control (Active Comparator): Participants in Group B will not receive any new interventions.
  Interventions: Other: No research related technology based social interactions

INTERVENTIONS:
Behavioral: Technology based social interactions — Participants will be socially interacting using any available technology with members of the research team.
  Arms: Group A Intervention
Other: No research related technology based social interactions — No technology based social interactions with the research team.
  Arms: Group B Control

SUMMARY:
The current study will examine the impact of frequent social interaction through communication technologies during COVID-19 pandemic in the cognitive status of socially-isolated older adults with and without cognitive impairment. Patients will take place in an experimental crossover study, participants will complete one month of an intervention and one month of as passive control. The goal of this study is to determine: A.) if frequent social interaction through ICT during COVID-19 pandemic will have a significant positive impact in cognitive performance on testing, and B.) how social isolation and cognitive status influence misconceptions around the current pandemic.

DETAILED DESCRIPTION:
The current study will examine the impact of frequent social interaction through communication technologies during COVID-19 pandemic in the cognitive status of socially-isolated older adults with and without cognitive impairment. An estimated 150 total participants will be recruited over the course of 1 year: 50 healthy older participants, 50 patients with amnestic mild cognitive impairment, and 50 patients with mild AD.

This study employs an AB/BA crossover design (2-sequence, 2-period, 2-treatment design) where A will be the intervention phase and B will be the passive control phase. Each period will occur over a duration of 1 month. Participants will either receive an intervention designed to provide participants with more social interaction during a time of social distancing and highly limited in-person social interactions (Intervention Group) or will not receive the intervention (Control Group). The investigators will conduct pre- and post- neuropsychological testing to assess changes in cognitive status (e.g., memory, language, executive functioning) in the intervention group after each intervention phase. Neuropsychological tests assessing changes to cognition will be completed prior to participant assignment to the Intervention or Control Group. Following this assessment, the first phase of the intervention will begin, and the initial intervention group (Group A) will receive the intervention, and the other group (Group B) will act as a control group. After the intervention phase has ended, both groups will be assessed again using neuropsychological tests. Following the re-assessment, Group B will receive the intervention, and Group A will act as a control. After the second intervention phase has ended, both groups will be assessed once more using neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis from the Boston University Alzheimer's Disease Center of mild AD (with a recent Mini Mental State Examination score greater than 20)
* Meet criteria for social isolation- a state in which an individual has a minimal number of social contacts and lacks engagement with others either physically or remotely through communication technology.
* English as their primary language
* Have access to either a computer, smart device, or telephone

Exclusion Criteria:

* Clinically significant depression
* Alcohol or drug use
* Cerebrovascular disease, traumatic brain damage, other degenerative disease (e.g., Parkinson's disease)
* Do not have corrected vision of 20/30 or better
* perform below 80% correct on the speech discrimination test from the Boston Diagnostic Aphasia Examination
* Score below 27 on the Mini-Mental State Examination (MMSE)
* Score below two standard deviations on any element of the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List Memory test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Change in memory performance | Baseline,1 month
  The Oral Trail Making Test B (TMT-B) will be used to assess memory performance. It is a neuropsychological measure that provides an assessment of sequential set-shifting. Participants are asked to count from 1 to 25 switching between number and letter, eg 1-A-2-B-3-C, until stopped.
Change in cognition | Baseline, 1 month
  Repeatable Battery for the Assessment of Neuropsychological Status (R-BANS) will be administered to assess cognitive decline or improvement. The 12 items on the RBANS assess five cognitive domains: immediate memory, visuospatial/constructional abilities, language, attention, and delayed memory. Scores can range from 0-160 and are interpreted as: 130 and above- very superior; 120-129 - superior; 110-119- high average; 90-109- average; 80-89- low average; 70-79- borderline; 60 and below extremely low.
Change in phonemic fluency | Baseline, 1 month
  Phonemic fluency will be assessed by asking participants to produce orally as many words as possible beginning with a specific letter or for a specific category (eg animals, fruits, etc). The test consists of three trials, of 1 min each. The higher the number of words provided, the greater the verbal fluency.

SECONDARY OUTCOMES:
Social isolation | 1 month
  The 6-item version of the Lubben Social Network scale (LSNS-6) will be used to assess social isolation. For each of the 6 questions the participant rates from 0 to 5 their perceived social engagement where 0=less social engagement and 5= more social engagement. The summed total score ranges between 0 and 30. Lower total scores indicate more social isolation.
Loneliness | 1 month
  Loneliness will be assessed using the UCLA loneliness scale. Participants rate each item as either O ("I often feel this way"= 3),S ("I sometimes feel this way"=2), R ("I rarely feel this way"=1), N ("I never feel this way"=0). A total score is computed by adding up the response to each question and can range from 0 to 60. The average loneliness score on the measure is 20. A score of 25 or higher reflects a high level of loneliness. A score of 30 or higher reflects a very high level of loneliness.
Depressive symptoms | 1 month
  The Geriatric Depression Scale (GDS) will be used to assess depression. It consists of 15 questions- 10 indicate the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicate depression when answered negatively. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Misinformation about Covid-19 | 1 month
  An investigator developed questionnaire based on survey results published by Geldsetzer P in Annals of Internal Medicine, 3-2020 will be used to assess Covid-19 misinformation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Busdon, MD, Principal Investigator — Professor of Neurology at BU School of Medicine
Locations (1):
- Boston University Alzheimer Disease Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vives-Rodriguez AL, Marin A, Schiloski KA, Hajos GP, Di Crosta A, Ceccato I, La Malva P, Anderson DC, Lahdo N, Donnelly K, Dong J, Kasha S, Rooney C, Dayaw J, Marton G, Wack A, Hanger V, DeCaro R, Di Domenico A, Turk KW, Palumbo R, Budson AE. Impact of remote social interaction during the COVID-19 pandemic on the cognitive and psychological status of older adults with and without cognitive impairment: A randomized controlled study. PLoS One. 2024 Nov 12;19(11):e0311792. doi: 10.1371/journal.pone.0311792. eCollection 2024. PMID 39531433